CLINICAL TRIAL: NCT06552624
Title: An Open-label, Randomized, Crossover Study to Investigate the Comparative Pharmacodynamics and Pharmacodynamics Equivalence of Antareit 800 Chewable Tablets and Riopan 800 mg Chewable Tablets in Healthy Volunteers
Brief Title: Comparative Pharmacodynamics and Pharmacodynamics Equivalence of Antareit 800 mg Chewable Tablets and Riopan 800 mg Chewable Tablets in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ANT-05-02-2021
Record Dates: First submitted 2024-07-19; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Heartburn; Acid-dependent Diseases of the Gastrointestinal Tract; Symptomatic Treatment of Gastric and Duodenal Ulcers
MeSH Terms: conditions — Heartburn; Duodenal Ulcer | interventions — magaldrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR-sequence (T-test drug, R-reference drug) (Experimental): Group 1 (20 volunteers, TR sequence) will take 2 tablets of Antareit (magaldrate) 800 mg chewable tablets 2 h prior to food intake in Period 1 and 2 tablets of Riopan (magaldrate) 800 mg chewable tablets 2 h prior to food intake in Period 2
  Interventions: Drug: Magaldrate
- RT-sequence (Experimental): Group 2 (20 volunteers, RT sequence) will take 2 tablets of Riopan (magaldrate) 800 mg chewable tablets 2 h prior to food intake in Period 1 and 2 tablets of Antareit (magaldrate) 800 mg chewable tablets 2 h prior to food intake in Period 2
  Interventions: Drug: Magaldrate

INTERVENTIONS:
Drug: Magaldrate — A dose of T drug in one of 2 periods of the study 2 h prior to food intake, 3 times per day
  Other Names: Antareit (T)
Drug: Magaldrate — A dose of R drug in one of 2 periods of the study 2 h prior to food intake, 3 times per day
  Other Names: Riopan (R)

SUMMARY:
Comparative study of the pharmacodynamic parameters and pharmacodynamic equivalence (bioequivalence) of drug Antareit 800 mg chewable tablets and drug Riopan 800 mg chewable tablets in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study prior to any of the study procedures;
2. Healthy male and female caucasian volunteers aged 18 to 45 years (inclusive);
3. Verified diagnosis "healthy" (without abnormal findings in the protocol-defined clinical, laboratory, and instrumental test data);
4. pH according to hourly pH-metry in the screening period, carried out at least 3 hours after the last meal, is completely in the range from 1 to 3 inclusive throughout the entire astronomical hour of measurement;
5. Blood pressure (BP) levels: 100 to 139 mm Hg, inclusive (systolic, SBP), 60 to 89 mm Hg, inclusive (diastolic, DBP);
6. Heart rate (HR) of 60 to 90 bpm, inclusive;
7. Body mass index (BMI) of 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2, where the body weight range is ≥ 55 kg for men and ≥ 45 kg for women;
8. Non-smoking healthy volunteers (who have never smoked or gave up smoking more than 6 months prior to the Screening);
9. Consent to use adequate methods of contraception throughout the study and for 30 days after completion; for women of preserved reproductive potential, a negative urine pregnancy test result;
10. The volunteers must have adequate behavior and coherent speech.

Exclusion Criteria:

1. A history of allergy;
2. History of drug intolerance to the active substance and/or excipients included in the study drugs;
3. History of drug intolerance of or hypersensitivity/allergic reactions to lidocaine, xylocaine or other topical anesthetics which will be used at the trial site for anesthesia during esophagogastroduodenoscopy (EGD) and insertion of the probe for the pH measurements;
4. Chronic diseases of the circulatory, lymphatic, respiratory, nervous, endocrine, gastrointestinal, musculoskeletal, integumentary, immune, urogenital, and hematopoietic systems;
5. Esophageal, gastric, and/or duodenal diseases based on EGD performed at screening and based on the medical history; a history of esophageal, gastric, and/or duodenal surgery;
6. Diseases/conditions which, in the opinion of the investigator, may affect the pH measurement results;
7. Acute infectious diseases less than 4 weeks prior to screening;
8. Use of antacids (including sodium bicarbonate solution)/H2 antagonists 24 h prior to the Screening Visit;
9. Use of proton pump inhibitors 72 h prior to the Screening Visit;
10. Use of (including use of a single dose) steroids and/or other ulcerogenic drug (e.g., nonsteriodal anti-inflammatory drugs [NSAID]) less than 4 weeks prior to the Screening Visit;
11. Regular use of any medicinal products, including prescription only and OTC (Over-the-counter) drugs and dietary supplements within 2 weeks prior to the Screening Visit;
12. Blood or plasma donation less than 3 months prior to the Screening Visit;
13. Use of hormonal contraceptives (in women) less than 2 months prior to the Screening Visit;
14. Pregnancy or breastfeeding; a positive pregnancy test for women of childbearing potential;
15. Participation in another clinical trial less than 3 months prior to screening or simultaneously with this study;
16. Use of more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 ml of beer, 150 ml of wine or 40 ml of spirits) a week within a month prior to the enrollment in the study or history data of alcohol/drug dependence or drug abuse.
17. Positive antibody blood test for HIV-1 and HIV-2, Treponema pallidum antigen, hepatitis B surface antigen (HBsAg), or hepatitis C virus antigen;
18. Positive urine test for narcotic substances or strong drugs;
19. Positive test for alcohol vapor in exhaled breath or a positive alcohol saliva test;
20. Deviated septum/nasal obstruction preventing the placement of the pH probe;
21. Medical history of chronic constipation;
22. Medical history of severe maxillofacial injuries;
23. Expected admission to hospital during this study for any reason, except for hospitalization provided for by this protocol;
24. Impossibility or failure to comply with the protocol, undergo protocol-defined procedures, or adhere to the diet or activity regime;
25. Other circumstances which in the opinion of the investigator prevent a volunteer from being included in the study or may result in premature drop-out from the study.

Withdrawal criteria:

1. The volunteer's refusal to further participate in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Taking prohibited therapy;
4. Occurrence of causes/occurrence during the study of situations that threaten the safety of the volunteer, including severe AEs;
5. Volunteers selected to participate in the study in violation of the inclusion/non-inclusion criteria;
6. Violation of the rules for conducting pH measurements or the occurrence of conditions that required early termination of pH measurements (vomiting, nosebleeds, etc.);
7. Missing a dose of the study drug/comparator drug during any period of the study for any reason;
8. Positive urine test for narcotics and strong drugs;
9. Positive breath alcohol vapor test or alcohol in saliva;
10. Positive pregnancy test in women;
11. The occurrence in the course of the study of other reasons that prevent the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics - AUCpH - Area under the curve potential of hydrogen above the baseline | From 0 to 1 hour (Day 1 and Day 8)
  Area under the pharmacodynamic pH-time curve adjusted to baseline (before drug intake)

SECONDARY OUTCOMES:
Pharmacodynamics - time percentage during which the intragastric pH value will exceed 4.0 | From 0 to 1 hour (Day 1 and Day 8)
  PH - potential of hydrogen
Pharmacodynamics - рН maximum | From 0 to 1 hour (Day 1 and Day 8)
  Maximum potential of hydrogen
Pharmacodynamics - рН minimum | From 0 to 1 hour (Day 1 and Day 8)
  Minimum potential of hydrogen
Pharmacodynamics - average pH value | From 0 to 1 hour (Day 1 and Day 8)
  Root mean square
Pharmacodynamics - time percentage during which the intragastric pH value will exceed 3.0 | From 0 to 1 hour (Day 1 and Day 8)
  Time during which the intragastric pH value will exceed 3.0
Pharmacodynamics - median time when the pH was above 3.0 | From 0 to 1 hour (Day 1 and Day 8)
  Time during which the intragastric pH value will be above 3.0
Pharmacodynamics - median time when the pH was above 4.0 | From 0 to 1 hour (Day 1 and Day 8)
  Time during which the intragastric pH value will be above 4.0
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: serious adverse event (SAE) number and frequency | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
  Number and frequency of serious AEs (SAEs)
Safety and Tolerability: volunteer complaints | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
  Description of complaints, recieved from volunteer
Safety and Tolerability: physical examination results - cardiovascular system | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the cardiovascular system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - respiratory system | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the respiratory system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - digestive tract | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the digestive tract on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - endocrine system | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the endocrine system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - musculoskeletal system | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the musculoskeletal system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - nervous system | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the nervous system on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - sensory systems | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the sensory systems on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: physical examination results - skin/visible mucous membranes | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  An assessment of the condition of the skin/visible mucous membranes on physical examination (normal condition or list of abnormal conditions, if any)
Safety and Tolerability: vital signs - systolic blood pressure | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  Systolic blood pressure (SBP, mmHg)
Safety and Tolerability: vital signs - diastolic blood pressure | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  Diastolic blood pressure (DBP, mmHg)
Safety and Tolerability: vital signs - heart rate | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  Heart rate (HR, bpm)
Safety and Tolerability: vital signs - body temperature (Celsius temperature scale) | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  Body temperature (Celsius temperature scale)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, Day 9
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, Day 9
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: PQ interval (is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, Day 9
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: QRS complex (the QRS complex is the combination of three of the graphical deflections seen on a typical electrocardiogram)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval | Screening, Day 9
  12-lead ECG (I, II, III, aVR-enhanced unipolar abduction from the right arm , aVL-enhanced unipolar abduction from the left arm, aVF - enhanced unipolar abduction from the left leg, V1-V6) taken while lying down: corrected QT interval (distance from the beginning of the QRS complex to the end of the T wave)
Safety and Tolerability: clinical blood test - hemoglobin | Screening, Day 2, Day 9
  Hemoglobin (g/L)
Safety and Tolerability: clinical blood test - hematocrit | Screening, Day 2, Day 9
  hematocrit (%)
Safety and Tolerability: clinical blood test - red blood cell count | Screening, Day 2, Day 9
  Red blood cell count (cells/L)
Safety and Tolerability: clinical blood test - platelet count | Screening, Day 2, Day 9
  Platelet count (cells/L)
Safety and Tolerability: clinical blood test - leukocyte count | Screening, Day 2, Day 9
  Leukocyte count (cells/L)
Safety and Tolerability: clinical blood test - erythrocyte sedimentation rate | Screening, Day 2, Day 9
  Erythrocyte sedimentation rate (m/h)
Safety and Tolerability: clinical blood test - myelocytes | Screening, Day 2, Day 9
  Leukocyte formula (myelocytes, %)
Safety and Tolerability: clinical blood test - band neutrophils | Screening, Day 2, Day 9
  Leukocyte formula (band neutrophils, %)
Safety and Tolerability: clinical blood test - segmented neutrophils | Screening, Day 2, Day 9
  Leukocyte formula (segmented neutrophils, %)
Safety and Tolerability: clinical blood test - eosinophils | Screening, Day 2, Day 9
  Leukocyte formula (eosinophils, %)
Safety and Tolerability: clinical blood test - basophils | Screening, Day 2, Day 9
  Leukocyte formula (basophils, %)
Safety and Tolerability: clinical blood test - monocytes | Screening, Day 2, Day 9
  Leukocyte formula (monocytes, %)
Safety and Tolerability: clinical blood test - lymphocytes | Screening, Day 2, Day 9
  Leukocyte formula (lymphocytes, %)
Safety and Tolerability: blood chemistry - glucose | Screening, Day 2, Day 9
  Glucose concentration (mmol/L)
Safety and Tolerability: blood chemistry - cholesterol | Screening, Day 2, Day 9
  Total cholesterol concentration (mmol/L)
Safety and Tolerability: blood chemistry - protein | Screening, Day 2, Day 9
  Total protein concentration (g/L)
Safety and Tolerability: blood chemistry - bilirubin | Screening, Day 2, Day 9
  Total bilirubin concentration (micromol/L)
Safety and Tolerability: blood chemistry - creatinine | Screening, Day 2, Day 9
  Creatinine concentration (micromol/L)
Safety and Tolerability: blood chemistry - alkaline phosphatase | Screening, Day 2, Day 9
  Alkaline phosphatase activity (U/L)
Safety and Tolerability: blood chemistry - alanine transaminase | Screening, Day 2, Day 9
  Alanine transaminase activity (U/L)
Safety and Tolerability: blood chemistry - aspartate transaminase | Screening, Day 2, Day 9
  Aspartate transaminase activity (U/L)
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 2, Day 9
  Specific gravity of the urine
Safety and Tolerability: urinalysis - color | Screening, Day 2, Day 9
  Color of the urine
Safety and Tolerability: urinalysis - transparency | Screening, Day 2, Day 9
  Transparency of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 2, Day 9
  pH of the urine
Safety and Tolerability: urinalysis - protein | Screening, Day 2, Day 9
  Protein concentration (g/L)
Safety and Tolerability: urinalysis - glucose | Screening, Day 2, Day 9
  Glucose concentration (mmol/L)
Safety and Tolerability: urinalysis - red blood cells | Screening, Day 2, Day 9
  Red blood cell content (number in sight)
Safety and Tolerability: urinalysis - white blood cells | Screening, Day 2, Day 9
  White blood cell content (number in sight)
Safety and Tolerability: urinalysis - epithelial cells | Screening, Day 2, Day 9
  Epithelial cell content (number in sight)
Safety and Tolerability: urinalysis - casts | Screening, Day 2, Day 9
  Presence of casts (Yes/No)
Safety and Tolerability: urinalysis - mucus | Screening, Day 2, Day 9
  Presence of mucus (Yes/No)
Safety and Tolerability: urinalysis - bacteria | Screening, Day 2, Day 9
  Presence of bacteria (Yes/No)
Safety and Tolerability: urinalysis (microscopy) | Screening, Day 2, Day 9
  Microscopy of urine sediment is performed if it is present

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Llc "Certa Clinic", Moscow
  - Private Health Care Institution "Clinical Hospital "RZD-Medicine" of St. Petersburg, Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided